CLINICAL TRIAL: NCT05093621
Title: Torsemide Comparison With Furosemide for Management of Patients With Stable Heart Failure
Acronym: TFO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000029589
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Torsemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Furosemide (Active Comparator): Furosemide, oral, dosage and frequency determined by treating physician or provider.
  1 mg torsemide to 2-4 mg oral furosemide
  Interventions: Drug: Furosemide
- Torsemide (Active Comparator): Torsemide, oral, dosage and frequency determined by treating physician or provider.
  1 mg torsemide to 2-4 mg oral furosemide
  Interventions: Drug: Torsemide

INTERVENTIONS:
Drug: Furosemide — Standard of care diuretic
  Arms: Furosemide
Drug: Torsemide — Standard of care diuretic
  Arms: Torsemide

SUMMARY:
The study is designed to be a prospective, randomized study is to compare the effectiveness of two standard of care loop diuretics (furosemide versus torsemide) on clinical outcomes among patients currently on a stable dose of loop diuretics.

DETAILED DESCRIPTION:
This study will be a randomized, unblinded, two-arm, multi-center clinical trial of patients receiving loop diuretics for treatment of heart failure in an outpatient clinic. This study will serve as additional enrollment for Cardio-Renal Effects of Torsemide vs. Furosemide: A TRANSFORMHF Mechanistic Sub-Study (HIC 2000025867) which is currently only enrolling patients admitted to the hospital for worsening heart failure. Thus allowing for expanded enrollment into HIC 2000025867 with a more diverse group of heart failure patients. Participants will be co-enrolled into this study and HIC 2000025867, NCT03296813.

Patients will be randomized 1:1 to either oral torsemide OR oral furosemide (dosing at discretion of local provider with dose equivalency guidance provided). This study will include stable subjects seen at the outpatient setting. The initial and follow-up dosing of torsemide and furosemide will be at healthcare provider discretion, with the following conversion provided as a guide: 1 mg torsemide to 2-4 mg oral furosemide. For instance, a patient would receive torsemide 20mg or furosemide 40-80 mg. Providers will be asked to document their planned initial dose and dosing frequency of torsemide and furosemide Randomization will occur within thirty days after the consent process and at the discretion of the healthcare provider and research team. Following randomization, the study medication is expected to constitute the oral diuretic therapy for one year. Patients will be prescribed the randomized study medication on the day of randomization.

Dose adjustments will be at the discretion of the treating healthcare provider(s) with strategies in place to maintain prescription of and adherence to the randomized medication. All patients will have 30-day, and 12-month post-randomization phone contacts for assessment of vital status, interval hospitalizations, concomitant HF medications, adherence, and weight.

To achieve these goals, the investigators propose a multi-center 125-patient study that will also co-enroll into Transform Ancillary (HIC 2000025867, NCT03296813) a mechanistic sub-study of this study and TRANSFORMHF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of heart failure and who have been on a stable dose of a diuretic for at least 30 days.
2. Plan for a daily outpatient oral loop diuretic regimen with anticipated need for long term loop diuretic use
3. ≥ 18 years of age
4. Signed informed consent

Exclusion Criteria:

1. End-stage renal disease requiring dialysis therapy
2. Inability or unwillingness to comply with the study requirements
3. History of heart transplant or actively listed for heart transplant
4. Implanted left ventricular assist device or implant anticipated <3 months
5. Pregnant or nursing women or women who are trying to conceive
6. Malignancy or other non-cardiac condition limiting life expectancy to <12 months
7. Known hypersensitivity to furosemide, torsemide, or related agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rao VS, Cox ZL, Ivey-Miranda JB, Neville D, Balkcom N, Moreno-Villagomez J, Ramos-Mastache D, Maulion C, Bellumkonda L, Tang WHW, Collins SP, Velazquez EJ, Mentz RJ, Wilson FP, Turner JM, Wilcox CS, Ellison DH, Fang JC, Testani JM. Mechanistic Differences between Torsemide and Furosemide. J Am Soc Nephrol. 2025 Jan 1;36(1):99-107. doi: 10.1681/ASN.0000000000000481. Epub 2024 Aug 28. PMID 39196651

RESULTS

PARTICIPANT FLOW:
Groups:
- Furosemide: Furosemide, oral, dosage and frequency determined by treating physician or provider.
  1 mg torsemide to 2-4 mg oral furosemide
  Furosemide: Standard of care diuretic
- Torsemide: Torsemide, oral, dosage and frequency determined by treating physician or provider.
  1 mg torsemide to 2-4 mg oral furosemide
  Torsemide: Standard of care diuretic
Period: Overall Study
Arm/Group | Furosemide | Torsemide
Started | 23 | 24
Yale Site Participants | 18 | 18
Completed | 23 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Furosemide | Torsemide | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (13.85) | 63.20 (12.05) | 61.93 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 15 | 19 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.87 (7.26) | 34.39 (9.13) | 34.13 (8.18)
Left ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: percentage of blood ejected] | 40.26 (14.94) | 43.40 (17.68) | 41.87 (16.26)
LVEF < 40% [Count of Participants; unit: Participants] — Number of participants with LVEF less than 40%
  Participants | 10 | 9 | 19
Ischemic cardiomyopathy [Count of Participants; unit: Participants] — Number of participants with Ischemic cardiomyopathy
  Participants | 7 | 7 | 14
Heart Failure hospitalization in the past year [Count of Participants; unit: Participants] | 4 | 4 | 8
Number of participants with comorbid conditions [Count of Participants; unit: Participants]
  Hypertension | 7 | 8 | 15
  Diabetes mellitus | 10 | 13 | 23
  History atrial fibrillation/flutter | 7 | 8 | 15
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 128.91 (16.07) | 127.62 (17.97) | 128.25 (16.89)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 77.43 (8.72) | 77.20 (10.10) | 77.31 (9.35)
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 66.86 (10.95) | 70.73 (9.31) | 68.80 (10.24)
Hypertension drugs [Count of Participants; unit: Participants] — Number of participants on Angiotensin-converting enzyme inhibitors (ACEi), Angiotensin II receptor blockers (ARB) or angiotensin receptor/neprilysin inhibitor (ARNI).
  Participants | 16 | 14 | 30
Beta blocker [Count of Participants; unit: Participants] | 23 | 20 | 43
Mineralocorticoid receptor antagonist [Count of Participants; unit: Participants] | 12 | 10 | 22
Daily Dose of prescribed heart medications [Median (Full Range); unit: milligrams] | 25 [12.5 to 25.0] | 25 [18.75 to 32.5] | 25 [12.5 to 32.5]
Sodium-glucose cotransporter-2 inhibitors (SGLT2i) [Count of Participants; unit: Participants] | 5 | 12 | 17
Hydralazine & Nitrates [Count of Participants; unit: Participants] | 1 | 1 | 2
Chronic oral loop diuretic dose in furosemide equivalents (mg) [Mean (Full Range); unit: milligrams furosemide equivalents] | 40 [20 to 40] | 40 [40 to 80] | 40 [20 to 80]
Thiazide [Count of Participants; unit: Participants] | 0 | 0 | 0
Serum sodium [Mean (Standard Deviation); unit: mmol/L] | 139.79 (2.59) | 139.86 (3.19) | 139.82 (2.87)
Serum chloride [Mean (Standard Deviation); unit: mmol/L] | 102.88 (2.76) | 101.66 (2.73) | 102.27 (2.78)
Serum potassium [Mean (Standard Deviation); unit: mmol/L] | 4.50 (0.46) | 4.69 (0.53) | 4.59 (0.5)
Serum bicarbonate [Mean (Standard Deviation); unit: mmol/L] | 21.53 (2.83) | 21.98 (3.43) | 21.76 (3.12)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.10 (0.43) | 1.21 (0.35) | 1.16 (0.39)
Blood urea nitrogen [Mean (Standard Deviation); unit: mg/dL] | 19.33 (9.66) | 23.54 (8.59) | 21.43 (9.29)
estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: ml/min/1.73 m^2] | 69.51 (23.13) | 58.84 (26.38) | 64.06 (25.16)
eGFR < 60 ml/min/1.73 m^2 [Count of Participants; unit: Participants] — Number of participants with eGFR less than 60 ml/min/1.73 m2
  Participants | 9 | 14 | 23
eGFR < 30 ml/min/1.73 m^2 [Count of Participants; unit: Participants] — Measure Description: Number of participants with eGFR less than 30 ml/min/1.73 m2
  Participants | 0 | 2 | 2
NT-pro-B-type natriuretic peptide [Mean (Full Range); unit: pg/ml] | 362.5 [108.25 to 1858.25] | 1550 [381 to 2583] | 883 [174 to 1888]
Hemoglobin [Mean (Standard Deviation); unit: g/dl] | 12.58 (2.16) | 13.59 (2.41) | 13.09 (2.32)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants All-cause Mortality, Measured at 1 Year.
Description: All-cause mortality as measured by phone calls at 30 days and 1 year
Time Frame: 30 days and one year
Population: Data presented here is from Yale site only. Only data from the Yale site was collected and analyzed. Data from other site could not be collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Torsemide
Number analyzed (Participants) | 18 | 18
Participants
  30 days | 0 | 0
  one year | 0 | 1
Statistical Analysis 1: Comparison: Furosemide vs Torsemide; Mortality at 1 year; Test type: Superiority; p = 1.000, t-test, 2 sided

2. Secondary Outcome: All-cause Hospitalization
Description: At least one hospitalization for any reason up to one year
Time Frame: up to one year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Torsemide
Number analyzed (Participants) | 18 | 18
Participants | 6 | 7
Statistical Analysis 1: Comparison: Furosemide vs Torsemide; Test type: Superiority; p = 0.729, t-test, 2 sided

3. Secondary Outcome: Total Hospitalizations
Description: Total number of hospitalizations total number of hospitalizations in one year
Time Frame: up to one year
Population: as for outcome 1
Measure: Mean (Full Range); unit: hospitalizations
Arm/Group | Furosemide | Torsemide
Number analyzed (Participants) | 18 | 18
hospitalizations | 0 [0 to 1] | 0 [0 to 4]
Statistical Analysis 1: Comparison: Furosemide vs Torsemide; Test type: Superiority; p = 0.650, t-test, 2 sided

4. Secondary Outcome: Change in Weight
Description: Change in weight up to one year
Time Frame: up to one year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Furosemide | Torsemide
Number analyzed (Participants) | 18 | 18
kilograms | -1.84 (4.9) | -3.04 (10.22)
Statistical Analysis 1: Comparison: Furosemide vs Torsemide; Test type: Superiority; p = 0.873, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: one year
Arm/Group | Furosemide | Torsemide
All-Cause Mortality (participants affected / at risk) | 0/23 | 1/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT05093621/Prot_SAP_000.pdf